CLINICAL TRIAL: NCT04970888
Title: Comparing the Effects of Combining Cognitive and Physical Exercise Training on Cognition, and Cerebral Blood Flow Regulation in Men and Women With Chronic Heart Failure
Acronym: ReCARDIO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); The Montreal Health Innovations Coordinating Center (MHICC) (Other)
Responsible Party: Principal Investigator, Louis Bherer, Associate scientific director, Direction of prevention, Montreal Heart Institute, Montreal Heart Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MP-33-2018-2406
Record Dates: First submitted 2021-07-12; First posted 2021-07-21 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Chronic Heart Failure; Aging
Keywords: cognition; physical exercise; cognitive training; brain functions; combined intervention; heart failure; biomarkers; cerebral vasoreactivity; fitness
MeSH Terms: conditions — Motor Activity; Heart Failure | interventions — Cognitive Training; Exercise

STUDY DESIGN:
Intervention Model Description: parallel assignment (1:1:1)
Who Masked: Investigator, Outcomes Assessor
Masking Description: This clinical trial is a single-blinded study. Research personnel performing the outcome assessments and investigators will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combined (Experimental): Combined physical exercise and cognitive training. The combined intervention will include a cognitive training with aerobic and resistance exercises training, three sessions per week for 6 months. Participants will be allowed to perform cognitive and exercise training sessions either home-based or centre-based.
  Interventions: Other: Cognitive training; Other: Exercise training; Other: Usual care
- Exercise (Experimental): The physical exercises intervention will include aerobic and resistance exercises training, three sessions per week for 6 months. Participants will be allowed to perform exercise training sessions either home-based or centre-based.
  Interventions: Other: Exercise training; Other: Usual care
- Usual care (Active Comparator): Usual medical care with no interventions
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Cognitive training — The cognitive training will involve attention control training and memory training, with thrice-weekly 30-min sessions.
  Two of these sessions will involve computer or tablet-based attentional control training targeting dual-tasking, updating and working memory, as well as inhibition and switching. Difficulty of cognitive training will be tailored to participants' performances. The remaining session will consist of memory training. Participants will be instructed mnemotechnic, as well as be taught about memory in aging in general.
  Arms: Combined
Other: Exercise training — Participants will follow a 20-week physical training program, with 60-min thrice-weekly trainings. The training sessions will start with a 5-min warm-up, followed by an aerobic training (20 min) after which 20-min of resistance/muscular training will take place. The program will end with a 10-min cool-down. Training will be adapted to individuals' baseline capacity as measured by the baseline cardiorespiratory test. For home-training sessions, participants will have access to a complete exercise training program. A certified kinesiologist will supervise trainings. With the Heart rate sensor Polar H10, all the characteristics of the activities will be recorded (type of the activity, intensity, heart rate, duration). A kinesiologist will call participants every week to ensure the smooth running of the exercises training sessions and individualize the care according to the patient's level.
  Arms: Combined; Exercise
Other: Usual care — All patients will receive usual care and be treated according to evidence-based treatments. This will include optimal medical therapy, systematic information regarding dietary and fluid management, and a recommendation for regular physical activity consistent with the latest update of the Canadian Cardiovascular Society Guidelines for the Management of Heart Failure. Moreover, patients who benefit from a prescription for a cardiovascular rehabilitation program will be able to follow it, but they will not receive other forms of intervention for the duration of the study.

SUMMARY:
The objective of this project is to assess the effects of combined physical exercise and cognitive training interventions on cognitive and brain health in patients with heart failure (HF). Also, the role of sex on the effects of the interventions will be assessed.

DETAILED DESCRIPTION:
Cognitive impairment (CI) affects up to 50% of patients with heart failure (HF), and is associated with high mortality rates, poor quality of life, reduced functional capacities, and an overwhelming economic burden in Western countries. Non-pharmacological strategies could help enhance cognition in HF patients with CI. Combined physical exercise and cognitive training interventions have recently shown promising enhancement effects on cognition in patients with cardiovascular risk factors and mild cognitive impairment. The effects of combined interventions have never been tested in HF.

The main objective is to assess the effects of combined physical exercise and cognitive training interventions on cognition in patients with HF. Secondary objectives include: to characterize baseline and intervention-related changes in cerebral autoregulation, pulsatility and neurovascular coupling and to assess the role of sex on intervention effects.

Two-hundred and sixteen participants (36 men and 36 women/group) with stable HF regardless of aetiology and LVEF will take part in this study. All participants will have signed a written consent form before taking part in the study.

Patients will be stratified according to sex and LVEF (FEVG < 40% et FEVG > 40%), and will be randomly assigned to one of the 3 following study arms: 1) Combined physical exercise and cognitive training; 2) Physical exercise alone; and 3) Usual medical care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years old
* Stable chronic HF on maximally tolerated background treatment for at least 2 months (stable therapy with ACE-I, ARBs and MRA for at least 2 months), regardless of LVEF
* with no limitation of physical activity in ordinary physical activity (i.e. NYHA class I), moderate symptoms (i.e. NYHA class II) or marked limitation in activity (i.e. NYHA class III)
* Able to perform cognitive and physical training.

Exclusion Criteria:

* Acute cardiovascular event 1 month prior to randomization, including emergency visit or hospitalization for decompensated HF, acute myocardial infarction, stroke, and transient ischemic attack
* Planned cardiovascular intervention within 6 months (implantation of any cardiac device, cardiac revascularization, heart transplantation)
* Severe exercise intolerance
* Contraindications for exercise testing (e.g., uncorrected severe aortic or carotid stenosis, severe pulmonary hypertension, severe non-revascularizable coronary disease including left main coronary stenosis, significant myocardial ischemia or arrhythmia during low-intensity exercise, acute HF)
* Severe respiratory disease
* Non-cardiopulmonary limitation to exercise (e.g., arthritis, claudication or any peripheral neurological disease including other neurodegenerative diseases such as disabling Parkinson)
* Uncontrolled diabetes or untreated thyroid dysfunction
* Current or recent malignancy with life expectancy < 1 year
* Chronic hemodialysis or peritoneal dialysis
* Unable to read the informed consent form or unable to understand the oral explanations provided by the assessor.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in general cognitive functioning | Baseline and post-intervention at 6 months
  Montreal Cognitive Assessment (0-30 score, with a higher score indicating a better cognitive functioning).
Change in processing speed | Baseline and post-intervention at 6 months
  Validated remote version of neuropsychological tests and iPad tests (Composite Z-score).
Change in executive functions | Baseline and post-intervention at 6 months
  Validated remote version of neuropsychological tests and iPad tests (Composite Z-score).
Change in episodic memory | Baseline and post-intervention at 6 months
  Validated remote version of neuropsychological tests (Composite Z-score).

SECONDARY OUTCOMES:
Change in cerebral autoregulation - frontal cortical region | Baseline and post-intervention at 6 months
  Variations of prefrontal cortical oxygen saturation (rSO2, [HbO]/([HbO]+[HbR])) will be measured by Near Infrared Spectroscopy (NIRS), as a surrogate of cortical blood flow. Variations of continuous peripheral blood pressure (mm Hg) will be simultaneously measured by plethysmography at the finger. Autoregulation indices (unitless) will be derived from the correlation between variations of oxygen saturation measures and variations of peripheral blood pressure.
Change in cerebral autoregulation - middle cerebral arteries | Baseline and post-intervention at 6 months
  Variations of cerebral blood flow velocity (cm/s) at the level of the middle cerebral artery will be measured by Transcranial Doppler (TCD). Variations of continuous peripheral blood pressure (mm Hg) will be simultaneously measured by plethysmography at the finger. Autoregulation indices (unitless) will be derived from the correlation between variations of cerebral blood flow measures and variations of peripheral blood pressure.
Change in cerebral pulsatility - cortical frontal region | Baseline and post-intervention at 6 months
  Pulsatility will be measured as the normalized difference of relative near-infrared light intensity changes between systole and diastole, using NIRS in the prefrontal cortical region.
Change in cerebral pulsatility - middle cerebral arteries | Baseline and post-intervention at 6 months
  Pulsatility will be measured as the normalized difference of relative blood flow velocities between systole and diastole, using TCD in the middle cerebral arteries
Change in cerebral activity | Baseline and post-intervention at 6 months
  Significant changes in brain activity evoked by a Stroop task relative to baseline will be assessed by t-statistics maps, computed from variations of [HbO] and [HbR] measured by NIRS at the prefrontal cortex.

OTHER OUTCOMES:
Change in cardiorespiratory fitness | Baseline and post-intervention at 6 months
  Maximum incremental cardiopulmonary exercise test (VO2 max (ml.kg.min)
Change in 6-min walking test performance | Baseline and post-intervention at 6 months
  maximum distance performed in 6 minutes (distance, m)
Change in upper limb muscle strength | Baseline and post-intervention at 6 months
  Grip strength test score (kg).
Change in quality of life | Baseline and post-intervention at 6 months
  score on the 23 items of the Kansas City Cardiomyopathy Questionnaire (KCCQ)
Change in perceived self care behaviour | Baseline and post-intervention at 6 months
  European Heart Failure Self-care Behaviour Scale (EHFScB-9) will be completed. This self-reported questionnaire assesses the adherence to different self-care behaviours (e.g., eating low-salt diet, etc.).
Change in anxiety | Baseline and post-intervention at 6 months
  State-Trait Anxiety Inventory questionnaire (Score ranges from 20-80, with a higher score indicating higher anxiety).
Change in depressive symptoms | Baseline and post-intervention at 6 months
  Geriatric Depression Scale questionnaire (Score ranges from 0-30, with a higher score indicating larger depressive symptomatology).
Change in sleep quality | Baseline and post-intervention at 6 months
  Pittsburgh Sleep Quality Index questionnaire (Score ranges from 0-21, with a higher score indicating worse sleep quality). symptomatology).
Cognitive reserve | Baseline
  Rami and colleagues' cognitive reserve questionnaire (Scale ranges from 0-26, with a higher score indicating a greater cognitive reserve).
Genotyping data | baseline
  genotyping data that include the APOE gene
Change in NT-pro-BNP | Baseline and post-intervention at 6 months
  NT-pro-BNP (ng/L)
Change in high-sensitive Troponin T | Baseline and post-intervention at 6 months
  hsTnT (ng/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Louis Bherer, PhD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Preventive medicine and physical activity centre (centre EPIC), Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No